CLINICAL TRIAL: NCT06306833
Title: Psychophysiological Biomarkers to Assess the Effectiveness of Surface EMG Biofeedback as an Alternative Therapy to Reduce Chronic Low Back Pain
Brief Title: The Surface EMG Biofeedback as an Alternative Therapy to Reduce Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amaila Fazal [afazal] (Other)
Collaborators: University of Karachi (Other)
Responsible Party: Sponsor-Investigator, Amaila Fazal [afazal], Research Associate, Advanced Education & Research Center
Organization: Advanced Education & Research Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLBP-sEMG-14022024
Record Dates: First submitted 2024-02-21; First posted 2024-03-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sEMG Biofeedback Intervention (Experimental): Participants in the intervention group will receive biofeedback surface EMG (sEMG) therapy as an alternative therapy to reduce chronic low back pain
  Interventions: Other: Surface Electromyography (sEMG) Biofeedback
- Control (No Intervention): Participants in the control group will receive usual care

INTERVENTIONS:
Other: Surface Electromyography (sEMG) Biofeedback — Biofeedback sEMG therapy through the use of virtual aids like digital therapeutics would help reduce chronic low back pain in patients by overcoming their psychophysiological manifestations. All participants in the intervention group will receive sEMG biofeedback as an alternative therapy.
  Arms: sEMG Biofeedback Intervention

SUMMARY:
The prevalence of chronic low back pain (CLBP) among the Pakistani population is reported to be as high as 78% leading towards different physiological and psychosocial alterations with the worst cases suffering from disabilities. CLBP is a multifactorial phenomenon in which age, gender, comorbidities, lifestyle conditions, profession, working hours, and different stressors play their roles in its causation. However, different therapeutic techniques have been determined to reduce CLBP. Thus, this study aimed to assess the effectiveness of the biofeedback surface EMG (sEMG) technique in reducing chronic low back pain among sufferers in the long run.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a multifaceted condition with a range of adversative sequelae including mental and physical disability, social issues, and increased healthcare utilization. CLBP is one of the leading worldwide health problems however it has a benign nature. It is now accountable for more years lived with disability (YLDs) than any other chronic health problem. Chronic low back pain caused 72 million YLDs in 2013 approximately which is 1.5 times greater than that of depression and twice as high as that of diabetes. Further, in 2013, around 615 million individuals globally were affected by disabling chronic low back pain. Additionally, chronic low back pain and its accompanying disability also have a major economic burden on the country. According to an estimation, between 5 to 10% of low back pain cases will develop chronic low back pain (CLBP), which is ultimately accountable for the increased cost of treatment, a high number of sick leaves, and individual suffering and also one of the leading cause for individuals seeking health care services. Disparagingly, the issue of CLBP is not well understood in developing countries like Pakistan, Sri Lanka, India, and Bangladesh, which are in the process of development and experiencing economic development and a double burden of diseases. The chronic low back pain prevalence in Southeast Asian countries is reported to be very high, for instance much higher than that reported in the Western world. The prevalence of CLBP in Bangladesh is 64% followed by Pakistan which has a 40% prevalence rate and Sri Lanka and India 36% and 19%, respectively. Previous research studies have focused on the documentation of factors that are termed "yellow flags" which induce, aggravate, and enhance pain and disability in chronic low back pain patients. Psychological and social factors are considered important contributing factors in the bio-psychosocial approach for chronic low back pain management and its relationship with disability. Moreover, this study is in line with the United Nations' Sustainable Developmental Goals (UN-SDG) 2030 plan; Goal 3.d i.e. to "strengthen the capacity of all countries, in particular developing countries, for early warning, risk reduction and management of national and global health risks". Thus, this study protocol will be a randomized controlled trial that is specifically designed to compare the biofeedback surface EMG effectiveness for chronic low back pain in the Pakistani population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who constantly experience low back pain for the last three months.
* Individuals who seek care from healthcare provider due to low back pain
* Individuals with average pain intensity, were assessed using the Brief Pain Inventory (BPI) over the past week ≥ 2 on a 0-10 scale.
* Individuals with an average Oswestry Disability Index (ODI) score ≥ 4.
* Individuals with State-Trait Anxiety Inventory (STAI) score ≥ 20.

Exclusion Criteria:

* Age below or above 25 and 75 years, respectively.
* Females who are pregnant, lactating, or that they anticipate becoming pregnant in the next 3-6 months will be excluded.
* Individuals having any diagnosed chronic disease.
* Individuals having any diagnosed neurological disorder including Alzheimer's, Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Parkinson's, Stroke
* Individuals having any diagnosed motor disorder or had pathologic fractures of the spine, avascular necrosis or osteonecrosis, severe osteoarthritis. Including a history of spine surgery or a hip arthroplasty
* Individuals with an active cancer
* Blind individuals
* Individuals having a body mass index greater than 35 kg/m2
* Individuals with clinical depression, that is having a score of 24 or higher on the Center for Epidemiology Depression Scale.
* Individuals who have used narcotics or muscle relaxants within 30 days before study enrollment.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity and interference | 3 Months
  The Brief Pain Inventory (BPI) will be used to assess the severity of chronic low back pain and its impact on lower back functioning. Participants will rate the pain severity and the degree of interference. Using a 0-10 scale, where 0-4 corresponds to mild pain, 5-6 corresponds to moderate pain, and 7-10 corresponds to severe pain
Lower back pain related Disability | 3 Months
  The Oswestry Disability Index (ODI) will be used to categorize the degree of disability in CLBP patients. Each section is scored on a 0-5 scale, where 5 represents the greatest disability. The index is calculated by dividing the summed score and expressed as a percentage. Where, 0 - 20 indicates mild disability, 20 - 40% indicates moderate disability, 40 - 60% indicates severe disability, 60 - 80% indicates disabling, and 80 - 100% indicates bedridden or functional impairment.
Quality of Life with chronic low back pain | 3 Months
  The quality of life questionnaire will be used to assess the patient's perspective of their life quality. The score can range from 6-112. A higher score indicates a higher quality of life, where, a score of 90 is the average for a healthy population
Pain and Disability-related Anxiety | 3 Months
  The State-Trait Anxiety Inventory-STAI will be used for anxiety screening. It is a 20-item scale with a score range of 20-80, where higher score indicate higher levels of anxiety symptoms

SECONDARY OUTCOMES:
Substance P | 3 Months
  Changes in the levels of Substance P will be observed during the span of the study in the control and intervention groups.
Cortisol | 3 Months
  Changes in the levels of Cortisol will be observed during the span of the study in the control and intervention groups.
Beta Endorphins | 3 Months
  Changes in the levels of Beta Endorphins will be observed during the span of the study in the control and intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shamoon Naushad, Study Chair — Advanced Education & Research Center
Locations (1):
- Psychophysiology Lab, University of Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tagliaferri SD, Miller CT, Owen PJ, Mitchell UH, Brisby H, Fitzgibbon B, Masse-Alarie H, Van Oosterwijck J, Belavy DL. Domains of Chronic Low Back Pain and Assessing Treatment Effectiveness: A Clinical Perspective. Pain Pract. 2020 Feb;20(2):211-225. doi: 10.1111/papr.12846. Epub 2019 Nov 11. PMID 31610090
- [Background] Global Burden of Disease Study 2013 Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 301 acute and chronic diseases and injuries in 188 countries, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Aug 22;386(9995):743-800. doi: 10.1016/S0140-6736(15)60692-4. Epub 2015 Jun 7. PMID 26063472
- [Background] Hoy D, Geere JA, Davatchi F, Meggitt B, Barrero LH. A time for action: Opportunities for preventing the growing burden and disability from musculoskeletal conditions in low- and middle-income countries. Best Pract Res Clin Rheumatol. 2014 Jun;28(3):377-93. doi: 10.1016/j.berh.2014.07.006. Epub 2014 Oct 22. PMID 25481422
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Gaskin DJ, Richard P. The economic costs of pain in the United States. J Pain. 2012 Aug;13(8):715-24. doi: 10.1016/j.jpain.2012.03.009. Epub 2012 May 16. PMID 22607834
- [Background] Sa KN, Moreira L, Baptista AF, Yeng LT, Teixeira MJ, Galhardoni R, de Andrade DC. Prevalence of chronic pain in developing countries: systematic review and meta-analysis. Pain Rep. 2019 Dec 6;4(6):e779. doi: 10.1097/PR9.0000000000000779. eCollection 2019 Nov-Dec. PMID 31984290
- [Background] Karran EL, Grant AR, Moseley GL. Low back pain and the social determinants of health: a systematic review and narrative synthesis. Pain. 2020 Nov;161(11):2476-2493. doi: 10.1097/j.pain.0000000000001944. PMID 32910100
- [Background] Khan MNU, Morrison NMV, Marshall PW. The Role of Fear-Avoidance Beliefs on Low Back Pain-Related Disability in a Developing Socioeconomic and Conservative Culture: A Cross-Sectional Study of a Pakistani Population. J Pain Res. 2020 Sep 23;13:2377-2387. doi: 10.2147/JPR.S258314. eCollection 2020. PMID 33061553
- [Background] Bishwajit G, Tang S, Yaya S, Feng Z. Participation in physical activity and back pain among an elderly population in South Asia. J Pain Res. 2017 Apr 15;10:905-913. doi: 10.2147/JPR.S133013. eCollection 2017. PMID 28450787
- [Background] Nicholas MK, Linton SJ, Watson PJ, Main CJ; "Decade of the Flags" Working Group. Early identification and management of psychological risk factors ("yellow flags") in patients with low back pain: a reappraisal. Phys Ther. 2011 May;91(5):737-53. doi: 10.2522/ptj.20100224. Epub 2011 Mar 30. PMID 21451099
- [Background] van Erp RMA, Huijnen IPJ, Jakobs MLG, Kleijnen J, Smeets RJEM. Effectiveness of Primary Care Interventions Using a Biopsychosocial Approach in Chronic Low Back Pain: A Systematic Review. Pain Pract. 2019 Feb;19(2):224-241. doi: 10.1111/papr.12735. Epub 2018 Dec 2. PMID 30290052
- [Background] Dwyer CP, MacNeela P, Durand H, O'Connor LL, Main CJ, McKenna-Plumley PE, Hamm RM, Reynolds B, Conneely S, Slattery BW, Taheny D, NicGabhainn S, Murphy AW, Kropmans T, McGuire BE. Effects of Biopsychosocial Education on the Clinical Judgments of Medical Students and GP Trainees Regarding Future Risk of Disability in Chronic Lower Back Pain: A Randomized Control Trial. Pain Med. 2020 May 1;21(5):939-950. doi: 10.1093/pm/pnz284. PMID 31846024